CLINICAL TRIAL: NCT05629689
Title: A Phase 1a/1b, Multi-Centre, Open-Label, Dose-Escalation and Dose-Expansion Study in Patients With Solid Tumour Malignancies to Evaluate GEH200520 Injection / GEH200521 (18F) Injection Safety and Tolerability, PET Imaging, Pharmacokinetics, and Changes in Imaging After Treatment
Brief Title: A Study to Evaluate GEH200520/GEH200521 (18F) Safety and Tolerability When Used for PET Scans in Patients With Solid Tumour Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-269-001; 2024-515218-42-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-11; First posted 2022-11-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Malignant Solid Tumor; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A Cohort 1 - 1 mg dose (Experimental): 1 mg mass dose of GEH200520 Injection with fixed dose of GEH200521 (18F) Injection administered together
  Interventions: Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part A; Diagnostic Test: Dynamic and Static - PET/CT scan
- Part A Cohort 2 - 2 mg dose (Experimental): 2 mg mass dose of GEH200520 Injection with fixed dose of GEH200521 (18F) Injection administered together
  Interventions: Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part A; Diagnostic Test: Dynamic and Static - PET/CT scan
- Part A Cohort 3 - 4 mg dose (Experimental): 4 mg mass dose of GEH200520 Injection with fixed dose of GEH200521 (18F) Injection administered together
  Interventions: Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part A; Diagnostic Test: Dynamic and Static - PET/CT scan
- Part A Cohort 4 - 8 mg dose (Experimental): 8 mg mass dose of GEH200520 Injection with fixed dose of GEH200521 (18F) Injection administered together
  Interventions: Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part A; Diagnostic Test: Dynamic and Static - PET/CT scan
- Part A Cohort 5 (optional) - 12 or 15 mg dose (Experimental): 12 or 15 mg mass dose of GEH200520 Injection with fixed dose of GEH200521 (18F) Injection administered together
  Interventions: Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part A; Diagnostic Test: Dynamic and Static - PET/CT scan
- Part A Cohort 6 - Optimal dose (Experimental): Selected (optimal) mass dose as determined from results of Cohorts 1 through 5 of GEH200520 Injection with fixed dose of GEH200521 (18F) Injection administered together
  Interventions: Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part A; Diagnostic Test: Dynamic and Static - PET/CT scan
- Part B (Experimental): Selected (optimal) dose of GEH200520 Injection from Part A with fixed dose of GEH200521 (18F) Injection administered together in 3 sequential repeat imaging visits
  Interventions: Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part B; Diagnostic Test: Static - PET/CT scan

INTERVENTIONS:
Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part A — Administration of GEH200520 Injection followed within 2 to 4 minutes by GEH200521 (18F) Injection followed by a 10mL saline flush
  Arms: Part A Cohort 1 - 1 mg dose; Part A Cohort 2 - 2 mg dose; Part A Cohort 3 - 4 mg dose; Part A Cohort 4 - 8 mg dose; Part A Cohort 5 (optional) - 12 or 15 mg dose; Part A Cohort 6 - Optimal dose
Diagnostic Test: Dynamic and Static - PET/CT scan — Dynamic whole-body PET/CT scan starting at the time of injection (sequential scans over 90 minutes anticipated) followed by static whole-body scans starting at 150 minutes, 270 minutes, and (optional) 24 hours after injection.
  Arms: Part A Cohort 1 - 1 mg dose; Part A Cohort 2 - 2 mg dose; Part A Cohort 3 - 4 mg dose; Part A Cohort 4 - 8 mg dose; Part A Cohort 5 (optional) - 12 or 15 mg dose; Part A Cohort 6 - Optimal dose
Drug: GEH200520 Injection / GEH200521 (18F) Injection - Part B — Administration of GEH200520 Injection followed within 2 to 4 minutes by GEH200521 (18F) Injection followed by a 10mL saline flush
  Arms: Part B
Diagnostic Test: Static - PET/CT scan — Whole-body PET/CT scan (up to 30 min). Exact timing will be determined from Part A. An optional dynamic scan may be acquired in addition to the required whole-body PET/CT scan at each imaging visit.
  Arms: Part B

SUMMARY:
Part A: The purpose of this part is to assess the safety of GEH200520 and GEH200521 (18F) when administered to patients with solid cancer. Subjects will be requested to complete 3 study visits: 1 screening visit, 1 imaging visit (over 24 hours) and 1 follow-up visit (7 days later). The estimated duration of Part A is 21 days.

Part B: The purpose of this part of the study is to assess the imaging quality and findings as well as the safety and tolerability of GEH200520 and GEH200521 (18F) when administered to patients with cancer before and after immunotherapy treatment.

Subjects will be requested to complete 7 study visits: 1 screening visit, the first imaging visit, followed by 2 immunotherapy immune-checkpoint inhibitor (ICI) treatment visits and 2 additional imaging and 1 follow-up visit. Two late imaging transfer expected post follow up visit. The estimated duration for subject participation in Part B is approximately 64 days.

ELIGIBILITY:
Inclusion Criteria:

* The subject is able and willing to comply with all study procedures as described in the protocol, including the imaging day pre-visit requirements, and has read, signed, and dated an informed consent form prior to any study procedures being performed.
* The subject is male or female, ≥18 years of age.
* Subject has a life expectancy ≥12 weeks.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Subject has an unresectable or metastatic solid tumour or a local and resectable head and neck squamous cell carcinoma, or an unresectable stage III-IV melanoma.
* Subject is eligible for ICI treatment per Investigator judgement.
* Subject has at least 1 measurable tumour lesion documented on CT/magnetic resonance imaging (MRI) RECIST v1.1 during the last 12 months.
* Subject has a tumour lesion(s) of which a biopsy can safely be obtained according to standard clinical care procedures.
* Subject is male or female that agrees to adhere to the protocol contraception methods.

Exclusion Criteria:

* Subject is unable to undergo all procedures in the study and/or is unable to remain still and tolerate the imaging procedure.
* Subject has 12-lead ECG significant findings during screening, per Investigator's assessment.
* Subject is not stable due to medical condition or therapy that, in the opinion of the Investigator, could compromise subject safety or protocol objectives.
* Subject has active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents.
* Subject has serious non-malignant disease or conditions that, in the opinion of the Investigator, could compromise subject safety or protocol objectives.
* Subject has B or T cell lymphoma.
* Subject has brain or bone-marrow metastasis that, in the opinion of the Investigator, could compromise subject safety or protocol objectives.
* Subject has signs or symptoms of systemic infection within 2 weeks prior to imaging day.
* Subject has history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanised antibodies or fusion proteins or known allergy to the study IMP ingredients and/or the proposed ICI therapy.
* Subject has any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the ICI treatment, or that may affect the interpretation of the results or render the subject at high risk from complications.
* Subject has laboratory values out of range per protocol.
* Subject has any safety laboratory test results (blood chemistry, haematology, and urinalysis) that, in the opinion of the Investigator, could compromise subject safety or protocol objectives.
* Subject has had any major surgery within 4 weeks prior to enrollment.
* Subject has been enrolled in another interventional clinical study within the 30 days before screening for this study, except for the study site IIS.
* Subject is pregnant or planning to become pregnant or is breastfeeding.
* Subject has a history of alcohol or drug abuse within the last year.
* Subject has had treatment with systemic immunostimulatory agents within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to dosing with the IMP.
* Subject has had treatment with systemic immunosuppressive medications within 2 weeks prior to dosing with the IMP.
* Subject has received acute, low-dose, systemic immunosuppressant medications that, in the opinion of the Investigator, could compromise protocol objectives.
* Subject has used systemic corticosteroids to treat inflammatory or autoimmune symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2029-03-10 (Estimated); Study Completion 2029-03-10 (Estimated)

PRIMARY OUTCOMES:
Part A: The incidence of AEs upon causality to the IMPs. | Part A: 7 days
Part A: The severity of AEs per National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) upon causality to the IMPs. | Part A: 7 days
To evaluate the time-course changes in GEH200521 (18F) Injection uptake after immune-checkpoint inhibitor (ICI) treatment cycles compared to baseline. | Part B: 50 days

SECONDARY OUTCOMES:
To evaluate the radiation dosimetry of a fixed dose of GEH200521 (18F) Injection when administered with the different GEH200520 Injection mass doses by cumulated activity in source regions and by entire body. | 7 days
To evaluate the optimal imaging time window for GEH200521 (18F) Injection positron emission tomography (PET) imaging when administered with different GEH200520 Injection mass doses for Part A subjects. | 7 days
To determine the appropriate mass dose of GEH200520 Injection for administration with GEH200521 (18F) Injection to achieve an acceptable PET image quality for Part A subjects. | 7 days
To characterize the pharmacokinetic (PK) properties (AUC) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection for Part A subjects. | 7 days
  The PK parameter to be assessed: AUC
To characterize the pharmacokinetic (PK) properties (Cmax) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection for Part A subjects. | 7 days
  The PK parameter to be assessed: Cmax
To characterize the pharmacokinetic (PK) properties (CL) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection for Part A subjects. | 7 days
  The PK parameter to be assessed: CL
To characterize the pharmacokinetic (PK) properties (V) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection for Part A subjects. | 7 days
  The PK parameter to be assessed: V
To characterize the pharmacokinetic (PK) properties (t1/2) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection for Part A subjects. | 7 days
  The PK parameter to be assessed: t1/2
Collection of the incidence, severity, changes between visits for AEs/SAEs/AESIs, for Part A subjects. | 7 days
  Incidence of AEs, SAEs, and Treatment-emergent AEs by system organ class and preferred term
Changes in physical examination status following administration of GEH200520 and GEH200521 (18F) for Part A subjects | Baseline, 24 hours, 7 days post IMP administration
  The findings in the physical exam pre and post-administration will be summarized.
Change from baseline in the results of serum biochemistry test results following administration of GEH200520 and GEH200521 (18F) for Part A subjects. | Baseline, 24 hours, 7 days post IMP administration
  In this context, baseline is defined as the pre-treatment assessment at the screening visit. The occurrence of post injection values outside of normal limits and changes from baseline will be summarized.
Change from baseline in the results of haematology test results following administration of GEH200520 and GEH200521 (18F) for Part A subjects. | Baseline, 24 hours, 7 days post IMP administration
  Change from baseline in the results of haematology test results following administration of GEH200520 and GEH200521 (18F) for Part A subjects.
Changes in heart rate as beats per minute following administration of GEH200520 and GEH200521 (18F) for Part A subjects | Baseline, 2 hours, 24 hours, 7 days post IMP administration
  The occurrence of post-administration heart rate values outside the normal limits will be summarized.
Changes in blood pressure in mmHg following administration of GEH200520 and GEH200521 (18F) for Part A subjects | Baseline, 2 hours, 24 hours, 7 days post IMP administration
  The occurrence of post-administration blood pressure values outside the normal limits will be summarized.
Changes in temperature as degree C following administration of GEH200520 and GEH200521 (18F) for Part A subjects | Baseline, 2 hours, 24 hours, 7 days post IMP administration
  The occurrence of post-administration body temperature values outside the normal limits will be summarized.
Change from baseline in the results of 12-lead electrocardiograms (ECGs) following administration of GEH200520 and GEH200521 (18F) for Part A subjects | Baseline, 2 hours, 24 hours, 7 days post IMP administration
  Descriptive statistics will be used to describe the observed values and change from baseline.
To assess immunogenicity, via the incidence of treatment-induced anti-drug antibodies responses, after a single injection of the different GEH200520 Injection mass doses administered with a fixed dose of GEH200521 (18F) Injection for Part A subjects. | 7 days
Collection of the incidence, severity, changes between visits for AEs/SAEs/AESIs | 50 days
To assess the biodistribution and tumour uptake of GEH200521 (18F) Injection with the optimal GEH200520 Injection dose determined in Part A based on quantitative measurements of GEH200521 (18F) in regions of interest for Part B subjects. | 50 days
To assess the relationship between tumour GEH200521 (18F) Injection uptake (SUV value) and immune cell CD8+ expression score from a biopsy sample/resected lesion when available based on IHC results for Part B subjects. | 50 days
To compare changes in tumour GEH200521 (18F) Injection uptake with changes in computed tomography (CT) image assessment, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 for Part B subjects when available . | 50 days
To compare changes in tumour GEH200521 (18F) Injection uptake with changes in computed tomography (CT) image assessment, according to [18F]-fluorodeoxyglucose (FDG) scans, when available for Part B subjects. | 50 days
Changes in physical examination status following administration of GEH200520 and GEH200521 (18F) for Part B subjects | Baseline, Day 15, Day 36, Day 50
  The occurrence of post-administration physical exam status values outside the normal limits will be summarized.
Change from baseline in the results of serum biochemistry test results following administration of GEH200520 and GEH200521 (18F) for Part B subjects. | Baseline, Day 15, Day 36, Day 50
  In this context, baseline is defined as the pre-treatment assessment at the screening visit. The occurrence of post injection values outside of normal limits and changes from baseline will be summarized.
Change from baseline in the results of haematology test results following administration of GEH200520 and GEH200521 (18F) for Part B subjects. | Baseline, Day 15, Day 36, Day 50
  In this context, baseline is defined as the pre-treatment assessment at the screening visit. The occurrence of post injection values outside of normal limits and changes from baseline will be summarized.
Changes in heart rate as beats per minute following administration of GEH200520 and GEH200521 (18F) for Part B subjects | Baseline, Day 15, Day 36, Day 50
  The occurrence of post-administration heart rate values outside the normal limits will be summarized.
Changes in blood pressure in mmHg following administration of GEH200520 and GEH200521 (18F) for Part B subjects | Baseline, Day 15, Day 36, Day 50
  The occurrence of post-administration blood pressure values outside the normal limits will be summarized.
Changes in temperature as degree C following administration of GEH200520 and GEH200521 (18F) for Part B subjects | Baseline, Day 15, Day 36, Day 50
  The occurrence of post-administration body temperature values outside the normal limits will be summarized.
Change from baseline in the results of 12-lead electrocardiograms (ECGs) following administration of GEH200520 and GEH200521 (18F) for Part B subjects | Baseline, Day 15, Day 36, Day 50
  Descriptive statistics will be used to describe the observed values and change from baseline.
To characterize the PK properties (AUC) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of GEH200520 Injection with GEH200521 (18F) Injection for Part B subjects. | 50 days
  The PK parameter to be assessed: AUC
To characterize the PK properties (Cmax) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of GEH200520 Injection with GEH200521 (18F) Injection for Part B subjects. | 50 days
  The PK parameter to be assessed: Cmax
To characterize the PK properties (CL) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of GEH200520 Injection with GEH200521 (18F) Injection for Part B subjects. | 50 days
  The PK parameter to be assessed: CL
To characterize the PK properties (V) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of GEH200520 Injection with GEH200521 (18F) Injection for Part B subjects. | 50 days
  The PK parameter to be assessed: V
To characterize the PK properties (t1/2) of total protein (GEH200520 and [18F]GEH200521 combined) following administration of GEH200520 Injection with GEH200521 (18F) Injection for Part B subjects. | 50 days
  The PK parameter to be assessed: t1/2
To compare immunogenicity, via the incidence of treatment-induced anti-drug antibodies responses, after multiple administrations of GEH200520 Injection with GEH200521 (18F) Injection for Part B subjects. | 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Raiter, MD, Study Director — GE Healthcare
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - UMC Groningen, Groningen